CLINICAL TRIAL: NCT00850668
Title: A Phase 1 Study of Heat/Phenol-Killed, E. Coli-Encapsulated, Recombinant Modified Peanut Proteins Ara h 1, Ara h 2, and Ara h 3 (EMP 123) in Healthy Volunteers Followed by Subjects Allergic to Peanuts (CoFAR 1)
Brief Title: Peanut Allergy Vaccine Study in Healthy and Peanut-allergic Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allertein Therapeutics, LLC (Industry)
Collaborators: Consortium of Food Allergy Research (Other)
Responsible Party: Sponsor
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CoFAR1; COFAR; APA-001
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Food Hypersensitivity; Hypersensitivity; Immediate Hypersensitivity; Peanut Hypersensitivity
Keywords: Food Allergy; Peanut Allergy
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity; Hypersensitivity, Immediate; Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMP-123 (Active Comparator): Participants who are not allergic to peanuts will receive four escalating doses of study product on a weekly basis
  Interventions: Biological: E. Coli-Encapsulated, Recombinant Modified Peanut Proteins Ara h 1, Ara h 2, and Ara h 3
- EMP-123 in Peanut Allergics (Experimental): Participants who are allergic to peanuts will receive weekly dose escalation of the study product for 10 weeks followed by administration every 2 weeks for 6 weeks
  Interventions: Biological: E. Coli-Encapsulated, Recombinant Modified Peanut Proteins Ara h 1, Ara h 2, and Ara h 3

INTERVENTIONS:
Biological: E. Coli-Encapsulated, Recombinant Modified Peanut Proteins Ara h 1, Ara h 2, and Ara h 3 — Up to 7 mL solution administered rectally
  Other Names: EMP-123

SUMMARY:
The purpose of this study is to evaluate the safety and side effects of a study product that contains recombinant modified peanut proteins (EMP-123) in healthy and peanut-allergic participants. This is a first in human study.

As of November 2009, this study is no longer recruiting healthy volunteers and will only be recruiting individuals with peanut allergies.

DETAILED DESCRIPTION:
Peanut allergy is a common ailment in the United States. Research suggests that the prevalence of peanut allergy in the United States has doubled over the last 5 years. Currently, the only effective treatment for peanut allergy is a peanut-free diet and quick access to self-injectable epinephrine. This study will evaluate the safety of a rectally administered product, EMP-123, consisting of three recombinant modified peanut protein antigens encapsulated within dead E. coli. E. coli is a common bacterium found in everyone's colon. E. coli acts like a package to hold the modified peanut proteins. EMP-123 is designed to act as an allergy vaccine with an eventual goal to induce tolerance to the major peanut proteins responsible for peanut allergy.

This study will involve weekly dosing and for females, a pregnancy test will occur at 48 hours before the start of product administration and later during the study. The study will involve two steps. Step 1 will enroll 5 healthy participants who will receive four escalating doses of study product on a weekly basis. Participants will be monitored at the clinic for 2 hours after receiving each dose of study product. Each dosing visit will be followed with a phone interview to assess any adverse effects or symptoms. Participants in Step 1 will maintain a home diary and record any symptoms that occur between visits. After screening, Step 1 will consist of five study visits on Weeks 1, 2, 3, 4, and 8. Vital signs, adverse event monitoring, and review of the home diary will occur at all visits. Breathing tests will occur at most visits. Stool and urine collection will occur at Weeks 4 and 8. The expected duration of Step 1 is 8 weeks.

If no safety concerns are identified at the conclusion of Step 1, 10 peanut-allergic participants will be enrolled into the second phase of the study, Step 2.

Step 2 is expected to last 20 weeks. Participants in Step 2 will receive weekly dose escalation of the study product for 10 weeks followed by administration every 2 weeks for 6 weeks. Participants will remain in the clinic for 2 hours after every dose is received. Follow-up will then continue for 4 weeks after the conclusion of treatment. Each dosing visit will be followed with a phone interview to assess any adverse effects or symptoms. After screening, Step 2 will consist of 14 study visits. Vital signs, adverse event monitoring, and a review of the home diary will occur at all visits. Breathing tests will occur at most visits. A skin prick test and stool, blood, and urine collection will occur at select visits.

As of November 2009, this study is no longer recruiting healthy volunteers and will only be recruiting individuals with peanut allergies.

ELIGIBILITY:
Inclusion Criteria:

* Available for the duration of the trial
* Ability to perform spirometry maneuvers
* Agree to use effective methods of contraception for the duration of the study
* For Step 1 participants, regular consumption of at least 5 grams of peanut at least twice per month during the last 6 months prior to study entry
* For Step 2 participants, a convincing clinical history of peanut allergy and prick skin test positive to peanut. More information on these criteria can be found in the protocol.

Exclusion Criteria:

* History of any severe anaphylaxis
* Known allergy to hydroxypropyl methylcellulose, glycerol, or phenol
* Evidence of clinically significant immunosuppressive neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease
* Laboratory evidence of liver or hematologic disease. Pre-existing history of autoimmune or antibody mediated diseases. More information on this criterion can be found in the protocol.
* Pre-existing history of autoimmune or antibody mediated diseases. More information on this criterion can be found in the protocol.
* Any previous intubation due to allergies or asthma
* History of ischemic cardiovascular disease
* Uncontrolled hypertension
* Significant medical condition that, in the opinion of the investigator, would interfere with the study
* Chronic diarrhea
* Inability to refrain from anal intercourse for the duration of the trial
* Use of rectal medications during the study
* Planned rectal procedures for the duration of the study
* History of rectal surgery or bleeding in the last 6 months prior to study entry
* History of proctitis in the last 6 months prior to study entry
* History of inflammatory bowel disease, celiac disease, or eosinophilic esophagitis/gastroenteritis
* Participation in another investigational vaccine or drug trial within 30 days prior to study or while the study is ongoing
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the last 12 months prior to study entry
* FEV1 value less than 80% predicted
* Inability to discontinue antihistamines for skin testing
* Currently on any allergy immunotherapy
* Participation in any interventional study for the treatment of food allergy in the past 12 months prior to study entry
* Poor control of persistent activation of atopic dermatitis
* Use of omalizumab or other non-traditional forms of allergen immunotherapy or immunomodulatory therapy or biologic therapy within the past 12 months prior to study entry
* Use of oral B-blockers, angiotensin-receptor blockers, or calcium channel blockers
* Use of immunosuppressive drugs within 30 days prior to study entry or while study is ongoing
* Use of corticosteroids within 30 days prior to study entry
* Use of steroid medications. More information on this criterion can be found in the protocol.
* History of serologic evidence of infection with HIV-1, HBV, or HCV
* Receipt of blood products within the past 6 months prior to study entry
* Inability to refrain from anal intercourse for the duration of the study
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, would interfere with the study
* Pregnant or breastfeeding

Step 1 participants:

* History of any allergy to food, including peanut
* Serum peanut-specific IgE greater than .35 kUa/L at screening
* Prick skin test (PST) to peanut more than 3mm in diameter at screening
* History of asthma

Step 2 participants:

* More than mild persistent asthma as defined in the protocol.
* Treatment for asthma, including: any hospitalization in the past year for asthma or any emergency room visit in the past 6 months for asthma.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who successfully complete the dosage regimen with no more than mild symptoms related to EMP-123 dosing | Throughout study

SECONDARY OUTCOMES:
Occurrence of adverse events | Throughout study
Rate of desensitization, as determined by peanut endpoint titration prick test in peanut allergic participants | At pre- and post-treatment periods
Change in basophil activation | Throughout study
Decreased Type 2 helper T cell peanut-induced T-lymphocyte phenotype and increased T-lymphocyte regulatory phenotype | Throughout study
Increase in peanut-specific immunoglobulin (IgG4) and IgA | Throughout study
Decrease in peanut-specific IgE | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Wood, MD, Study Chair — Johns Hopkins University; Scott Sicherer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York

REFERENCES:
- [Background] Rolland JM, Gardner LM, O'Hehir RE. Allergen-related approaches to immunotherapy. Pharmacol Ther. 2009 Mar;121(3):273-84. doi: 10.1016/j.pharmthera.2008.11.007. Epub 2008 Dec 7. PMID 19111571
- [Background] Sicherer SH, Sampson HA. Peanut allergy: emerging concepts and approaches for an apparent epidemic. J Allergy Clin Immunol. 2007 Sep;120(3):491-503; quiz 504-5. doi: 10.1016/j.jaci.2007.07.015. Epub 2007 Aug 8. PMID 17689596